CLINICAL TRIAL: NCT03674840
Title: Comparison of Optical Quality With Different Placement of Refractive Multifocal Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hong Qi, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180906
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Cataract, Age-Related
Keywords: Multifocal Intraocular Lenses; visual acuity; kappa angle
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Parallel Assignment. For each patient one eye was randomly selected as design group and receive a SBL-3 implantation based on angle kappa, while the other eye was included in control group and receive a SBL-3implantation of 0 to 180 degree
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Subjects in this group will go through a cataract surgery with SBL-3 implantation in the direction of 0 to 180 degree guided by Callisto Eye System(Carl Zeiss Meditec, Germany) intraoperatively.
  Interventions: Procedure: 0 to 180 degree SBL-3 implantation
- design group (Experimental): Subjects in this group will go through a cataract surgery with SBL-3 implantation based on kappa angle(described by Pentacam HR preoperatively) guided by Callisto Eye System(Carl Zeiss Meditec, Germany) intraoperatively.
  Interventions: Procedure: angle kappa based SBL-3 implantation

INTERVENTIONS:
Procedure: angle kappa based SBL-3 implantation — SBL-3 implantation based on kappa angle guided by Callisto Eye System(Carl Zeiss Meditec, Germany) intraoperatively.
  Arms: design group
Procedure: 0 to 180 degree SBL-3 implantation — SBL-3 implantation in the direction of 0 to 180 degree guided by Callisto Eye System(Carl Zeiss Meditec, Germany) intraoperatively.
  Arms: control group

SUMMARY:
The study aims to compare postoperative optical quality between two different implanting position of a rotationally asymmetric MIOL [SBL-3 Lenstec; +3.00 diopters (D)], angle kappa based implantation and 0 to 180 degree implantation, in order to find out the optimal implantation position for SBL-3.

DETAILED DESCRIPTION:
SBL-3 has been proved to provide patients with good near, intermediate and distant visual acuity, but there is not much study on the impact of SBL-3 position on postoperative visual acuity.The regional refractive design of SBL-3 means it could be affected by pupil center shift (described by angle kappa: the difference between visual axis and pupil axis), the investigators assume that maintaining the ideal ratio of distant and near segment(50% vs 42%) in the pupil center could yield both good distant and near postoperative visual acuity postoperatively. Therefore, the investigators designed the implantation by placing the IOL based on angle kappa to make sure the ratio of distant and near segment exposure in the pupil center close to 50:42. In this study, the investigators assessed the optical quality in patients with SBL-3 implantation based on angle kappa and 0 to 180 degree to provide surgeons with information for choosing appropriate implantation position for optimum postoperative satisfaction of SBL-3.

ELIGIBILITY:
Inclusion Criteria:

* age related cataract
* underwent bilateral cataract surgery and SBL-3 implantation
* corneal astigmatism <1.5D

Exclusion Criteria:

* patients with active ocular inflammation
* neuro-ophthalmic disease and macular disease
* previous corneal or intraocular surgery, corneal opacities or disease
* patients had surgical complications, pupillary trauma, inability to place the lens in the capsular bag
* IOL tilt or decentration deviated from intraoperative positioning
* difficulties with examinations and follow-up

Ages: 54 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected visual acuity | 3 months postoperatively
  Comparison of uncorrected distance visual acuity (UCVA), intermediate visual acuity, near visual acuity were measured at 5m, 80cm and 33cm respectively. All visual acuity measurements were conducted under photopic conditions (85 cd/m2) and at 100% contrast in design group and control group.

SECONDARY OUTCOMES:
Optical quality | 3 months postoperatively
  An OPD scan III aberrometer (NIDEK Co. Ltd., Gamagori, Japan) was used to evaluate postoperative mesopic and photopic pupil diameters and the quality of vision in each subject. Visual acuity was evaluated by MTF(modulation transfer function), SR(strehl ratio), intraocular total aberration, high order aberration, spherical aberration, coma aberration, trefoil aberration under 4mm pupil diameter.
Contrast sensitivity | 3 months postoperatively
  Contrast sensitivity measures were conducted uniocularly, under photopic, mesopic (5 cd/m2), photopic with glare and mesopic with glare conditions, with the OPTEC 6500 contrast sensitivity test (Stereo Optical, USA). Contrast sensitivity was evaluated at five spatial frequencies (1.5, 3, 6, 12, and 18 cycles per degree [cpd]). Patients were allowed 5 minutes to adapt to each illumination level before testing.
Defocus curve | 3 months postoperatively
  Monocular defocus curves were obtained in all patients, positioned at 5m under photopic (>85 cd/m 2 ) condition to measure the visual acuity with each defocus lens, representing the consecutive visual function of each eye. Negative lenses were added in 0.50 D steps and the visual acuity was recorded for each type of defocus level. The procedure was then repeated but with positive lenses. The range of defocus evaluated was from -4.00D to +2.00D.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China